CLINICAL TRIAL: NCT05049330
Title: Development and Testing of a Pediatric Cervical Spine Injury Risk Assessment Tool
Acronym: C-Spine
Status: Recruiting | Type: Observational
Sponsor: Julie Leonard (Other)
Responsible Party: Sponsor-Investigator, Julie Leonard, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: 5R01HD091347 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Cervical Spine Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation Cohort: The derivation cohort collected data to derive the clinical decision rule.
- Validation Cohort: The validation cohort collected data to validate the clinical decision rule

SUMMARY:
Cervical spine injuries (CSI) are serious, but rare events in children. Spinal precautions (rigid cervical collar and immobilization on a longboard) in the prehospital setting may be beneficial for children with CSI, but are poorly studied. In contrast, spinal precautions for pediatric trauma patients without CSI are common and may be associated with harm. Spinal precautions result in well-documented adverse physical and physiological sequelae. Of substantial concern is that the mere presence of prehospital spinal precautions may lead to a cascade of events that results in the increased use of inappropriate radiographic testing in the emergency department (ED) to evaluate children for CSI and thus an unnecessary, increased exposure to ionizing radiation and lifetime risk of cancer. Most children who receive spinal precautions and/or are imaged for potential CSI, and particularly those imaged with computed tomography (CT), are exposed to potential harm with no demonstrable benefit. Therefore, there is an urgent need to develop a Pediatric CSI Risk Assessment Tool that can be used in the prehospital and ED settings to reduce the number of children who receive prehospital spinal precautions inappropriately and are imaged unnecessarily while identifying all children who are truly at risk for CSI.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17 years
* Known or suspected exposure to blunt trauma

At least one of the following applies to the patient:

* Undergoing trauma team evaluation
* Transported from the scene to participating facility by EMS
* Undergoing cervical spine imaging at participating facility
* Transferred to participating facility with cervical spine imaging

Exclusion Criteria:

* Exposed to solely penetrating trauma (e.g. a gunshot or stab wound)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 0-17 years with known or suspected blunt trauma exposure that arrive at participating children's hospitals and meet study eligibility criteria. No exclusion based on sex/gender, race, ethnic group, or language.
Sampling Method: Non-Probability Sample
Enrollment: 22222 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Develop the Pediatric CSI Risk Assessment Tool in children with blunt trauma using prospective observational data obtained from ED providers | 8/1/2018 - 7/31/2022
Validate the Pediatric CSI Risk Assessment Tool in a separate population of children with blunt trauma using prospective observational data obtained from ED providers | 8/1/2020-7/31/2023

SECONDARY OUTCOMES:
Validate the Pediatric CSI Risk Assessment Tool using prospective observational data obtained from EMS providers. | 8/1/2018-7/31/2023

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, Oakland, California
  - Children's Hospital UC Davis Health, Sacramento, California
  - Children's Hospital Colorado, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leonard JC, Harding M, Cook LJ, Leonard JR, Adelgais KM, Ahmad FA, Browne LR, Burger RK, Chaudhari PP, Corwin DJ, Glomb NW, Lee LK, Owusu-Ansah S, Riney LC, Rogers AJ, Rubalcava DM, Sapien RE, Szadkowski MA, Tzimenatos L, Ward CE, Yen K, Kuppermann N. PECARN prediction rule for cervical spine imaging of children presenting to the emergency department with blunt trauma: a multicentre prospective observational study. Lancet Child Adolesc Health. 2024 Jul;8(7):482-490. doi: 10.1016/S2352-4642(24)00104-4. Epub 2024 Jun 4. PMID 38843852
- [Derived] Tavender E, Eapen N, Wang J, Rausa VC, Babl FE, Phillips N. Triage tools for detecting cervical spine injury in paediatric trauma patients. Cochrane Database Syst Rev. 2024 Mar 22;3(3):CD011686. doi: 10.1002/14651858.CD011686.pub3. PMID 38517085

DOCUMENTS (4):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT05049330/Prot_000.pdf
  • Informed Consent Form: User Centered Design Cover Letter (2021-08-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT05049330/ICF_001.pdf
  • Informed Consent Form: CSI Identified Diversity Supplement Cover Letter (2021-08-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT05049330/ICF_002.pdf
  • Informed Consent Form: Consent Authorization Cover Letter (2021-08-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT05049330/ICF_003.pdf